CLINICAL TRIAL: NCT02228018
Title: The Comparison of Electronic Auscultation Coupled With Computer Aided Lung Sound Analysis (CALSA) and Functional Respiratory Imaging (FRI) and Repeatability of FRI Biomarkers in Healthy Subjects and Asthma Patients
Brief Title: The Comparison of Electronic Auscultation Coupled With CALSA and FRI; Repeatability of FRI Biomarkers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Other strategies followed
Sponsor: FLUIDDA nv (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLUI-2014-118
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CALSA and FRI repeatability (Experimental): CT-Scan No medication used
  Interventions: Device: CT-scan

INTERVENTIONS:
Device: CT-scan — CT-Scan will be taken at visit 1 on FRC and TLC breathing levels

SUMMARY:
CALSA will be compared with FRI and the repeatability of the FRI parameters will be tested in a group of healthy volunteers and asthma patients.

DETAILED DESCRIPTION:
his is a study with no investigational product. CALSA will be compared with FRI and the repeatability of the FRI parameters will be tested in a group of healthy volunteers and asthma patients.

Electronic auscultation of respiratory sounds will be performed, lung function tests (at maximal dilatation) will be executed and computed tomography (CT) scans of the thorax will be taken. The scans will be taken at two different breathing levels, more specifically at total lung capacity (TLC) and functional residual capacity (FRC) level. The scans will be taken while the patient/ volunteer lies down on the movable table of the CT-scan. After the scan is taken it will be asked to the patient/ volunteer to sit upright on the scanning table and to lie down again. When the patient/ volunteer lies down a second CT-scan (TLC and FRC) will be taken.

The objective of this study is to compare CALSA with FRI and to assess the repeatability of FRI biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient / volunteer ≥ 18 years old
* Written informed consent obtained
* The subject belongs to 1 of the following groups in the opinion of the investigator:

Group 1: healthy volunteer Group 2: patient with asthma

* Only if patient/ volunteer is a female of childbearing potential: Confirmation that a contraception method was used at least 14 days before visit 1

Exclusion Criteria:

* Pregnant or lactating female
* Patient/ volunteer with an uncontrolled disease or any condition that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study.

Patient/ volunteer with an uncontrolled disease or any condition that might, in the judgement of the investigator, place the patient at undue risk or potentially compromise the results or interpretation of the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
CALSA | 1 day
  The primary objective of this study is to compare CALSA with FRI. The respiratory sounds recordings are performed with a digital stethoscope and connected to the sound card of a laptop with commercial software, suitable for data acquisition. The respiratory sounds recordings are conducted in accordance with the Computerized Respiratory Sound Analysis guidelines (CORSA) for short-term acquisition. Subjects are asked to breathe through the mouth in a sitting position (tidal breathing) during the recordings. Three sets of recordings are made for 7 - 10 respiratory cycles with a maximum duration of 25 seconds.

SECONDARY OUTCOMES:
Total Airway Volume (iVaw) | 1 day
  The secondary objective is to check the repeatability of the FRI parameters
Total Airway Resistance (iRaw) | 1 day
  The secondary objective is to check the repeatability of the FRI parameters.
Internal Airway Distribution | 1 day
  The secondary objective is to check the repeatability of the FRI parameters
Lobar Volume | 1 day
  The secondary objective is to check the repeatability of the FRI parameters

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No